CLINICAL TRIAL: NCT03378115
Title: Energy Cost of Posture Maintenance, Ethnic Differences and the Influence of Metabolic State
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Other Study IDs: 2017/00285
Record Dates: First submitted 2017-12-15; First posted 2017-12-19 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Energy Expenditure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the magnitude of changes in energy expenditure and respiratory quotient (RQ) during sitting and standing in Asian men.

DETAILED DESCRIPTION:
The study will recruit 30-40 young healthy Asian men of Chinese, Malay or Indian descent. Volunteers will visit Clinical Nutrition Research Centre (CNRC) on 1 or 2 occasions: once for consenting and screening procedures (visit 1) and once to follow a 3 hour test session (visit 2). Consenting, screening and the test protocol can take place on the same day or can be scheduled on separate days. In this study the investigators will study the changes in energy expenditure and substrate oxidation when changing posture between sitting and standing. Visit 1 (screening): For screening, potential subjects will come in the morning after an overnight fast. After obtaining informed consent, a series of screening tests will be conducted, including questionnaires (general health, physical activity and eating behaviour), anthropometry (height, weight), blood pressure, resting heart rate, body composition and body proportions (waist circumference, hip circumference, sitting height, leg length, relative leg length, mid-arm circumference, mid-thigh circumference, calf circumference). The physical activity questionnaire will quantify physical activity level. The eating behaviour questionnaire will determine intentional restriction of food intake. Body composition will be measured using an electrical impedance analyser and the BodPod. Body proportions will be measured using a non-stretch measuring tape. Blood pressure and resting heart rate will be measured using an automatic blood pressure monitor. All these methods are non-invasive and do not cause any pain. Visit 2: This test session will last for approximately 3 hours in the morning, during which the following will take place: During each test session, the subject arrive at the centre between 8:00 and 9:00 in the morning after an overnight fast and has been instructed to avoid any physical activity/exercise and alcohol on the day prior to the test. The session will start after the subject enter the whole body calorimeter. The first 45 minutes after entering, resting metabolic rate will be measured. Therefore, the subject will lie down comfortably on a bed in a supine position. Over the following 60 minutes the subject will alternate a sitting and standing position every 15 minutes based on the researchers instructions. The subject will then receive a drink and snack to consume and there will be a 15 minute break in which the subject can take a toilet break if necessary. The break will be followed by a second sequence of 60 minutes in which the subject alternates a sitting and standing position every 15 minutes. After this subject will leave the whole body calorimeter and is free to go home.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male
* Age between 21-40 years old
* Chinese, Malay or Indian Ethnicity
* Body mass index between 18.5 - 28 kg/m2
* Normal blood pressure (<140/90 mmHg)
* Do not have metabolic diseases (such as diabetes, hypertension etc.)
* Do not have glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Do not take prescription medication that may affect metabolism
* Do not intentionally restrict food intake
* Do not have intolerances or allergies to test foods

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy males volunteers only
Study Population: Healthy Chinese/Malay/Indian
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Measurement of energy expenditure and respiratory quotient (RQ) in sitting and standing positions | Up to 3 hours
  Measured using Whole Body Calorimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Cenre, Singapore, Singapore

REFERENCES:
- [Derived] Camps SG, Koh HR, Henry CJ. Posture economy: the importance of metabolic state on metabolic phenotype assessment and the energy cost of sitting and standing. A whole body calorimetry trial. Eur J Clin Nutr. 2022 Aug;76(8):1178-1185. doi: 10.1038/s41430-022-01077-7. Epub 2022 Feb 1. PMID 35105942